CLINICAL TRIAL: NCT01722747
Title: Promoting Tobacco Control Among Teachers in India
Brief Title: Bihar School Teachers Study
Acronym: BSTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Healis-Sekhsaria Institute for Public Health (Other); Carelon Research (Other); University of Minnesota (Other); School of Preventive Oncology (Unknown)
Responsible Party: Principal Investigator, Glorian Sorensen, Professor of Society, Human Development and Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CA120958 (NIH)
Record Dates: First submitted 2012-11-01; First posted 2012-11-07 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Tobacco Use Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Condition (Experimental): Tobacco Free Teachers, Tobacco Free Society (TFT/TFS)
  Interventions: Behavioral: Tobacco Free Teachers, Tobacco Free Society (TFT/TFS)
- Delayed Intervention Control condition (No Intervention): Receives abbreviated 3-month delayed intervention after final data collection time point

INTERVENTIONS:
Behavioral: Tobacco Free Teachers, Tobacco Free Society (TFT/TFS) — A 7-month intervention was conducted over one academic year & included the following core components: 1. A Lead Teacher (LT) in each school was appointed and trained to facilitate the program on-site; 2. A tobacco policy was implemented; 3. Study health educators and LTs conducted group discussions with teachers addressing 6 intervention themes; 4. Materials; 5. Support for tobacco use cessation. Schools randomized to delayed intervention control condition did not receive any intervention until after final data collection, when they were given a 3-month shortened intervention.
  Arms: Intervention Condition

SUMMARY:
BRIEF SUMMARY: This study, which is closed to enrollment, is testing the efficacy of a tobacco-control intervention geared towards school teachers in Bihar, India. This cluster randomized trial aims to promote tobacco use cessation among teachers and increase tobacco policy adoption in 72 Bihar schools. Teachers are the focus of the study because as role models for youth and key opinion leaders related to community norms, they represent an important group for tobacco control. Teachers in Bihar also have reported high rates of tobacco use. According to the Global School Personnel Survey conducted in 2006, 39% of teachers in the eastern region of India (which includes Bihar) use some form of tobacco, compared to the national average of 29%. This study aims to reduce these numbers through discussion groups with teachers, individual cessation counseling, educational materials, and a tobacco policy workgroup in each intervention school. This study is a collaboration between US researchers and researchers at the Healis-Sekhsaria Institute for Public Health, Mumbai India.

ELIGIBILITY:
Inclusion Criteria:

* Government schools including grades 8-10 from within 10 school districts

Exclusion Criteria:

* Schools with fewer than 8 teachers
* Schools located in flood zones

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 945 (Actual)
Dates: Start 2009-06; Primary Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
6-month abstinence from tobacco | assessed 9-months post-intervention

SECONDARY OUTCOMES:
Adoption of a school tobacco policy | 9-month post-intervention
short-term tobacco use cessation | Average of 3 weeks post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Glorian C. Sorensen, PhD, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- School of Preventive Oncology, Patna, Bihar, India

REFERENCES:
- [Background] Nagler EM, Pednekar MS, Viswanath K, Sinha DN, Aghi MB, Pischke CR, Ebbeling CB, Lando HA, Gupta PC, Sorensen GC. Designing in the social context: using the social contextual model of health behavior change to develop a tobacco control intervention for teachers in India. Health Educ Res. 2013 Feb;28(1):113-29. doi: 10.1093/her/cys060. Epub 2012 Jun 4. PMID 22669010
- [Background] Pischke CR, Galarce EM, Nagler E, Aghi M, Sorensen G, Gupta PC, Pednekar MS, Sinha DN, Viswanath K. Message formats and their influence on perceived risks of tobacco use: a pilot formative research project in India. Health Educ Res. 2013 Apr;28(2):326-38. doi: 10.1093/her/cys112. Epub 2012 Dec 6. PMID 23221589